CLINICAL TRIAL: NCT00397332
Title: An Investigator Initiated Open-label and Explorative Study of Alefacept Treatment for Chronic Extensive Graft Versus Host Disease
Brief Title: Alefacept for Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Michael Shapira, MD, Hadassah University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYS-05-HMO-CTIL
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2011-02

CONDITIONS: Resistant Chronic GVHD
Keywords: GVHD
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alefacept — IM Alefacept

SUMMARY:
Alefacept (AMEVIVE®) is an immunosuppressive dimeric fusion protein that consists of the extracellular CD2-binding portion of the human leukocyte function antigen-3 (LFA-3) linked to the Fcof IgG1. Alefacept is produced by recombinant DNA technology in a Chinese Hamster Ovary (CHO) mammalian cell expression system. It was shown to interfere with lymphocyte activation. Alefacept was evaluated in two randomized, double-blind, placebo-controlled studies in adults with chronic plaque psoriasis. Each course consisted of once-weekly administration for 12 weeks of placebo or alefacept. The response to alefacept was significantly better in both studies. In both studies, onset of response to alefacept treatment (defined as at least 50% reduction of baseline Psoriasis Area and Severity Index (PASI)) began 60 days after the start of therapy. With one course of therapy, the median duration of response (defined as maintenance of a 75% or greater reduction in PASI) was 3.5 months for alefacept treated patients and 1 month for placebo-treated patients. Most patients who had responded to either alefacept or placebo maintained a 50% or greater reduction in PASI through the 3-month observation period.

Graft versus host disease (GVHD) is the most ominous side effect of allogenic stem cell transplantation (SCT). It causes severe inflammatory process, which is usually located to the skin, gut and liver. Treatment of GVHD consists of various immuno-suppressive and immuno-modulating drugs, including steroids, cyclosporine, tacrolimus, methotrexate etc. These drugs unfortunately can also cause severe immunologic failure that makes the patient prone to infection and malignancy, and other medication-specific side effects. In spite of this effect on the immune system, not all of the patients achieve control of GVHD, which usually rapidly leads to death. Despite the use of innovative immunosuppressive modalities, the prognosis of steroid resistant GVHD is usually poor. In the following study we will evaluate the effect of alefacept on steroid unresponsive cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* No age limit
* Resistant chronic GVHD

Exclusion Criteria:

* Not fulfilling any of the inclusion criteria
* Active life-threatening infection
* Inability to comply with study requirements.
* Known hypersensitivity to alefacept.
* Active malignant disease

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
GVHD response. | 6m
Time to GVHD response | 6m

SECONDARY OUTCOMES:
Overall survival. | 6m
Disease free survival. | 6m
Occurrence of infections. | 6m

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Department of Stem cell Transplantation & Cancer immunotherapy; Cell Therapy & Transplantation Biology Research Laboratory, Hadassah University Hospital
Locations (1):
- Department of Stem cell Transplantation & Cancer immunotherapy; Cell Therapy & Transplantation Biology Research Laboratory, Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Shapira MY, Resnick IB, Bitan M, Ackerstein A, Tsirigotis P, Gesundheit B, Zilberman I, Miron S, Leubovic A, Slavin S, Or R. Rapid response to alefacept given to patients with steroid resistant or steroid dependent acute graft-versus-host disease: a preliminary report. Bone Marrow Transplant. 2005 Dec;36(12):1097-101. doi: 10.1038/sj.bmt.1705185. PMID 16247429